CLINICAL TRIAL: NCT06936813
Title: Patients' and Physicians' Perspectives on the Management of Prolactinomas: Experiences, Treatment Preferences, and Related Outcomes - The PROMISE Survey
Brief Title: The PROMISE Survey
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00327; kt25Atila2
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prolactinoma; Pituitary Tumor
Keywords: Survey
MeSH Terms: conditions — Prolactinoma; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PROMISE Survey was developed to systematically assess the real-world experiences, treatment preferences, side effects, and outcomes from both patients and physicians dealing with prolactinomas. The aim is to generate insights that can guide future clinical research and improve individualized care strategies.

DETAILED DESCRIPTION:
Background

Prolactinomas are the most common hormone-producing pituitary tumors, causing symptoms like menstrual irregularities, infertility, galactorrhea, and reduced libido due to elevated prolactin levels. The standard treatment involves dopamine agonists (DAs) such as cabergoline or bromocriptine, which are usually effective. However, many patients report side effects (e.g., nausea, dizziness, psychiatric symptoms), leading to challenges in long-term adherence and uncertainty about outcomes after discontinuing therapy. Surgical treatment has emerged as a potentially safe and effective alternative, especially for selected patients, but perspectives from both patients and physicians on treatment preferences and outcomes are not well studied.

The survey is designed to be completed in 5-10 minutes, fostering high participation across diverse patient and physician populations. Data are collected anonymous covers the following areas:

1. Patient Characteristics
2. DA Therapy
3. Surgical Treatment
4. Diagnostic Pathway
5. Treatment Side Effects & Recurrence
6. Quality of Life and Psychosocial Impact
7. Physician Perspectives
8. Knowledge Gaps
9. Hypothesis Generation

Outcome

The collected data will inform:

* Better understanding of real-world management and challenges in prolactinoma care.
* Insights for improving clinical guidelines, patient education, and treatment decision-making.
* Hypotheses for future studies comparing outcomes of DA therapy vs. surgery and optimizing long-term management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Prolactinoma patients
* Prolactinoma treating physicians including endocrinologists and neurosurgeons

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Prolactinoma patients and physicians involved in the management of prolactinomas. Survey will be accessible globally via online patient communities, pituitary disorder organizations, physician networks, and in-clinic distribution.
Sampling Method: Probability Sample
Enrollment: 530 (Actual)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Generate hypotheses for future research | 6 months
  Generate real-world patient-centered data to identify patterns in treatment outcomes, patient-reported challenges, and areas where additional clinical trials are needed to develop new hypothesis for future research

SECONDARY OUTCOMES:
Collect data on patient characteristics | 6 months
  Distribution of patient demographics, cause of prolactinoma, additional pituitary disfunctions, symptom burden before diagnosis
Assess patient experiences with dopamine agonist (DA) therapy | 6 months
  Distribution of DA types and dosing, side effects, remission
Evaluate patient experiences with surgical treatment | 6 months
  Percentage of patients who underwent surgery, rate of complications, remission, additional treatment
Collect data on diagnostic pathways | 6 months
  Proportion of patients who underwent MRI or biochemical testing, number of consultations before diagnosis
Evaluate patient-reported quality of life (QoL) and psychosocial impact | 6 months
  Quality of life (QoL) and employment or lifestyle limitations due to symptoms or medication side effects, psychological comorbidities
Assess physician perspectives on treatment strategies | 6 months
  Distribution of first-line treatment preferences, criteria used for surgical referral, long-term monitoring, management strategies of endocrinologists and neurosurgeons
Investigate patient and physician knowledge gaps | 6 months
  Awareness of alternative treatment options, concerns about recurrence risk after therapy discontinuation, fertility and pregnancy management, patient satisfaction with treatment-related education and counseling

CONTACTS AND LOCATIONS:
Overall Officials: Cihan Atila, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland